CLINICAL TRIAL: NCT06692140
Title: Randomized Comparison of an Ultra-low Strut Thickness Everolimus-eluting Biodegradable Polymer Stent Versus Durable Polymer Everolimus-eluting Stents in Patients Treated with Percutaneous Coronary Intervention in an All Comer Population (The SORT OUT XII Trial)
Brief Title: Comparison of an Ultra-low Strut Thickness Everolimus-eluting Biodegradable Polymer Stent Versus Durable Polymer Everolimus-eluting Stents in Patients Treated with Percutaneous Coronary Intervention
Acronym: SORT OUT XII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SORT OUT XII STENT; VMK2401000 (Other: Odense University Hospital)
Record Dates: First submitted 2024-11-12; First posted 2024-11-18 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Ischemia, Myocardial; Coronary Artery Disease; Percutaneous Coronary Intervention (PCI)
Keywords: Drug-eluting stent; outcome
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Ultra-low strut thickness everolimus-eluting biodegradable polymer Evermine50 stent (Experimental): Percutaneous coronary interventin with Ultra-low strut thickness everolimus-eluting biodegradable polymer Evermine50 stent
  Interventions: Device: Ultra-low strut thickness everolimus-eluting biodegradable polymer Evermine50 stent(s)
- Everolimus-eluting stents (durable polymer everolimus-eluting Xience or Promus stent) (Active Comparator): Percutaneous coronary intervention with Everolimus-eluting stents (durable polymer everolimus-eluting Xience or Promus stent)
  Interventions: Device: PCI with Everolimus-eluting stents (durable polymer everolimus-eluting Xience or Promus stent(s))

INTERVENTIONS:
Device: Ultra-low strut thickness everolimus-eluting biodegradable polymer Evermine50 stent(s) — Percutaneous coronary intervention with Ultra-low strut thickness everolimus-eluting biodegradable polymer Evermine50 stent(s)
  Arms: Ultra-low strut thickness everolimus-eluting biodegradable polymer Evermine50 stent
Device: PCI with Everolimus-eluting stents (durable polymer everolimus-eluting Xience or Promus stent(s)) — Percutaneous coronary intervention with Everolimus-eluting stents (durable polymer everolimus-eluting Xience or Promus stent(s))
  Arms: Everolimus-eluting stents (durable polymer everolimus-eluting Xience or Promus stent)

SUMMARY:
The objective of this randomized study is to compare the safety and efficacy of the ultra-low strut thickness everolimus-eluting biodegradable polymer Evermine50 stent to the everolimus-eluting family stents (durable polymer everolimus-eluting Xience or Promus stents) in a population-based setting with coronary artery stenosis treated with percutaneous coronary intervention

ELIGIBILITY:
Inclusion Criteria:

* All patients aged ≥18 years who are eligible for treatment with one or several drug-eluting coronary stents

Exclusion Criteria:

* Age < 18 years
* Not able to consent to study participating (eg. intubated patients)
* Unstable circuit or in cardiogenic shock and therefore not able to understand the information and purpose of the study
* Do not speak Danish
* Already included in the SORT OUT XII study
* Life expectancy <1 year
* Allergic to study related treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3150 (Estimated)
Dates: Start 2024-11-16 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2032-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with target lesion failure | 1 year
  Target lesion failure (TLF) is a composite of cardiac death, myocardial infarction (not clearly attributable to a non-intervention lesion) or target lesion revascularization with percutaneous coronary intervention or coronary artery bypass operation

SECONDARY OUTCOMES:
Number of patients with all-cause death | 1 year, 3 years and 5 years
  All-cause death is defined as any death
Number of patients with cardiac death | 1 year, 3 years and 5 years
  Cardiac death is defined as death resulting from cardiovascular causes: death caused by acute myocardial infarction, death caused by sudden cardiac, including unwitnessed, death, death resulting from heart failure, death caused by cardiovascular procedures. Undetermined cause of death is defined as a death not attributable to any other category because of the absence of any relevant source documents. Such deaths will be classified as cardiovascular for end point determination
Number of patients with myocardial infarction | 1 year, 3 years and 5 years
  Myocardial infarction diagnosis follows "The Joint ESC/ACCF/AHA/WHF Task Force on "Third Universal Definition of acute myocardial infarction",which has been adapted by Academy Research Consortium. Acute myocardial infarction not related to other than index lesion is defined as any acute myocardial infarction that is not clearly attributable to a non-target vessel
Number of patients with definite stent thrombosis | 1 year, 3 years and 5 years
  Definite stent thrombosis is defined as:
  Angiographic confirmation of stent thrombosis. The presence of a thrombus that originates in the stent or in the segment 5 mm proximal or distal to the stent or in a side branch originating from the stented segment and the presence of at least one of the following criteria:
  Acute onset of ischemic symptoms at rest New electrocardiographic changes suggestive of acute ischemia Typical rise and fall in cardiac biomarkers (refer to definition of spontaneous myocardial infarction) Or Pathological confirmation of stent thrombosis
Number of patients with probable stent thrombosis | 1 year, 3 years and 5 years
  Probable stent thrombosis is defined as any myocardial infarction that is related to documented acute ischemia in the territory of the implanted stent without angiographic confirmation of stent thrombosis and in the absence of any other obvious cause regardless of the time after the index procedure,
Number of patients with target lesion revascularization | 1 year, 3 years and 5 years
  Target lesion revascularization is defined as a repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. The target lesion is defined as the treated segment including the 5-mm margin proximal and distal to the stent
Number of patients with target vessel revascularization | 1 year, 3 years and 5 years
  Target vessel revascularization is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel including the target lesion. The target vessel is defined as the entire major intervened coronary vessel, including side branches

CONTACTS AND LOCATIONS:
Overall Officials: Lisette O Jensen, Principal Investigator — Odense University Hospital
Locations (3):
- Denmark (3):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication
Supporting Information: Study Protocol
Time Frame: 12. NOV 2024 til the end of the study
Access Criteria: On request
URL: https://www.clinicaltrials.gov/